CLINICAL TRIAL: NCT06333795
Title: Faecal Microbiota Transplantation Against Chronic Diarrhea in Patients With Systemic Sclerosis - a Randomized, Double-blinded, Safety and Pilot-efficacy Study
Brief Title: Faecal Microbiota Transplantation Against Chronic Diarrhea in Patients With Systemic Sclerosis
Acronym: FaeMiCue
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Klaus Krogh, MD, DMSc, PhD, Professor, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-10-72-131-23
Record Dates: First submitted 2024-03-05; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Diarrhea; Systemic Sclerosis
Keywords: Faecal Microbiota Transplantation (FMT); Diarrhea; Systemic Sclerosis; Chronic Diarrhea
MeSH Terms: conditions — Diarrhea; Scleroderma, Systemic | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Participants will undergo 2 interventions. For the first intervention participants are randomised 1:1 for either Active FMT or placebo For the second intervention, all participants receive active treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is blinded throughout the active study period, both the patient and investigator are blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental): Active capsule FMT-treatment
  Interventions: Procedure: Faecal Microbiota Transplantation (FMT)
- Placebo (Placebo Comparator): Placebo capsules are given.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Faecal Microbiota Transplantation (FMT) — Treatment is given as capsules.
  Arms: Active treatment
Procedure: Placebo — Treatment is given as capsules.
  Arms: Placebo

SUMMARY:
This clinical trial aims to assess the safety and effectiveness of faecal Microbiota Transplantation (FMT) in improving chronic diarrhea symptoms among patients with systemic sclerosis.

DETAILED DESCRIPTION:
The present study aims to assess the feasibility, pilot efficacy, and safety of FMT for patients with Systemic Sclerosis.

Participants will undergo two interventions in this present study.

In the first intervention, participants are randomized 1:1 for either active FMT or Placebo. This first intervention consists of two doses of FMT with a 3-7 day gap.

In the second intervention, all participants receive 1 dose of active FMT treatment.

This study design allows researchers to evaluate the safety of FMT in this patient group, and compare the effects of FMT in the FMT-treated group vs the placebo group, to see if FMT promotes remission of Chronic diarrhea. Furthermore, researchers will be able to gain insights into whether 2 initial doses are superior to one.

ELIGIBILITY:
Inclusion Criteria:

* Participants > 18 years
* Fulfilling and previously diagnosed with SSc according to the 2013 American College of Rheumatology/European League against rheumatisms SSs classification criteria[23] by rheumatologist or dermatologist.
* Chronic diarrea is defined as loose or watery stools, three or more times a day, a minimum of 50% of the days within the last four weeks.

Exclusion Criteria:

* Inability to understand Danish spoken or written and/or Trial procedures.
* Known or anticipated pregnancy (excluded by male sex, postmenopausal women, or otherwise negative U-HCG)
* Previous treatment with FMT
* Treatment with antibiotics within the past 6 weeks
* Changes in morphine treatment within the past 4 weeks
* Ongoing infection with Clostridioides difficile (negative PCR test)
* Known serious gastrointestinal disease or GI infection (diagnosed with e.g. inflammatory bowel disease and/or gastrointestinal cancer)
* Dysregulated thyroid disease (TSH) blood sample from previous consultations maximum 6 months old from
* Known intestinal stricture
* Planned MR scan within the study period
* Pacemaker/ICD
* Previous abdominal surgery (minor surgical procedures ex. appendectomy is allowed)
* Changes in medicine that affect the GI tract within the past four weeks.
* Known Severe end-organ disease

  * Lung disease with forced vital capacity(FVC)<50% and/or diffusing lung capacity for carbon monoxide (DLCO) <40%
  * Severe heart failure with ejection fraction <30%
  * End-stage kidney disease with glomeration rate<30ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events (AE) severity grade 2 or more assessed by CTCAE v5.0. during the first week after intervention (FMT or placebo). | The first week after treatment.
  Patient-reported measures from the schedule of side effects and telephone call 1 week after each intervention.

SECONDARY OUTCOMES:
Patient-reported treatment outcome on symptoms | The first week after treatment.
  Based on self-reported data from the bowel habit diary.
Patient-reported measures from the schedule of side effects and telephone call 1 week after each intervention. | One week after each treatment
  Mild adverse events (grade 1) following FMT or placebo assessed by (Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0) CTCAE v5.0.
  The CTCAE grades adverse events (AEs) based on severity:
  Grade 1: Mild, asymptomatic, or mild symptoms; no intervention needed. Grade 2: Moderate; requires minimal intervention; affects age-appropriate activities.
  Grade 3: Severe or medically significant, not immediately life-threatening; may require hospitalization.
  Grade 4: Life-threatening; urgent intervention needed. Grade 5: AE-related death. Note: Some AEs may not have all five grades available.
Patient-reported outcomes from questionnaires. | At Baseline and 4 weeks after Intervention 1 & 2
  Change in Gastrointestinal syndrome rating scale - irritable bowel version questionnaire (GSRS-IBS)
Patient-reported outcomes from questionnaires. | At Baseline and 4 weeks after Intervention 1 & 2
  Change in Wexner incontinence score.
Patient-reported outcomes from questionnaires. | At Baseline and 4 weeks after Intervention 1 & 2
  Change in UCLA Scleroderma Clinical Trial Consortium Gastrointestinal Tract (UCLA SCTC GIT 2.0)
Patient-reported overall symptom burden | Each week for a total of 26 weeks.
  The patients self-reported the severity of symptoms and their impact on daily life each week on a scale from 1-5. 1 being little to no burden, 5 being most severe.
Objective measures from the wireless motility capsule. | At baseline
  Transit time through the small intestine.
Objective measures from the wireless motility capsule. | At baseline
  Colonic transit times
Objective measures from the wireless motility capsule. | At baseline
  Total gastrointestinal transittimes
Objective measures from the wireless motility capsule. | At baseline
  Ph drop from the small intestine to the colon
Objective measures from the low-dose CT scan. | At baseline and 4 weeks after first intervention
  Volume of the a) small intestine and b) the colon. Volume of gas in a) the small intestine and b) the colon.
  Changes in the gas volume in the small intestine and colon.
Breath Test | At baseline and 4 weeks after first intervention
  Changes in the rise of hydrogen and methane measured in breath test
Faecal microbiota composition | At baseline and between each treatment, up to 4 weeks after last intervention
  Changes in faecal microbiome composition. Alfa and beta diversity determined by sequencing of the intestinal microbiome.
Faecal-calprotectin | At Baseline and 4 weeks after Intervention 1 & 2
  Percentual change in faecal-calprotectin from before intervention to 4 weeks after each intervention.
Blood plasma proteomics | At baseline and between each treatment, up to four weeks after last intervention.
  Changes in blood immunological parameters (including proteins) from baseline and between each treatment, at 4 weeks after intervention.
Blood plasma Fibrosis markers | At baseline and between each treatment, up to four weeks after last intervention.
  Changes in blood immunological parameters (including markers of fibrosis) from baseline and between each treatment, at 4 weeks after intervention.
Blood parameters | At baseline and between each treatment, up to four weeks after last intervention.
  Changes in blood immunological parameters (including circulating cytokines) from baseline and between each treatment, at 4 weeks after intervention.
Health-related Quality of life | At baseline and 4 weeks after Intervention 1 & 2
  Changes in Health-related Quality of life assessed with (EQ-5D-5L). Each of the five dimensions comprising the EQ-5D descriptive system is divided into five levels of perceived problems: LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/Extreme problems
  An EQ-VAS from 0-100 is added, 100 being the best possible health.
Patient perception of FMT treatment satisfaction | At 4 weeks after interventions 1 & 2
  Patient perception of FMT treatment satisfaction was assessed by 7-point Likert scale for patients. 1: no benefits from treatment to 7 being very satisfied with treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark